CLINICAL TRIAL: NCT02987556
Title: Crossover Evaluation of the Safety and the Efficacy of Artificial Pancreas Diabeloop for Three Months at Home in Comparison With Conventional Treatment by External Insulin Pump in Patients With Type 1 Diabetes.
Brief Title: Diabeloop WP7 : Crossover Evaluation of the Safety and the Efficacy of Artificial Pancreas Diabeloop (WP7)
Acronym: WP7
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre d'Etudes et de Recherche pour l'Intensification du Traitement du Diabète (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2016-A01198-43
Record Dates: First submitted 2016-11-28; First posted 2016-12-09 (Estimated); Last update posted 2019-02-01 (Actual); Status verified 2018-05

CONDITIONS: Closed Loop; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Intervention Model Description: Closed loop vs. Open loop,
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual System (open-loop) (Active Comparator): In open loop, patients will be provided with an Continuous Glucose Monitoring (CGM) and an external insulin pump programmed with its usual treatment previously prescribed by its physician.
  Interventions: Device: Continuous Glucose Monitoring; Device: External Insulin Pump
- DIABELOOP System (closed-loop) (Experimental): In the closed-loop, patients will be provided with the Diabeloop system consisting of insulin pump Cellnovo or Kaleido driven by remote control augmented by Diabeloop software and connected to the CGM Prescription of insulin doses proposed by a predictive algorithm.
  Interventions: Device: Continuous Glucose Monitoring; Device: External Insulin Pump; Other: telemdecine; Device: The Diabeloop Software (Model predictive control)

INTERVENTIONS:
Device: Continuous Glucose Monitoring — Collection of glucose data
Device: External Insulin Pump — insulin delivery
Other: telemdecine — Remote follow up by care health providers team
  Arms: DIABELOOP System (closed-loop)
Device: The Diabeloop Software (Model predictive control) — Diabeloop is a Closed-loop (CL) system with a Model Predictive Control (MPC) algorithm reinforced by a decisional matrix, uploaded on a dedicated android smartphone linked to Dexcom CGM and a Cellnovo or Kaleido insulin patch-pump. The Diabeloop software calculates the insulin dose according to the patient's needs.
  Arms: DIABELOOP System (closed-loop)

SUMMARY:
The study will be conducted in crossover trial, with two 12-weeks periods separated by a Wash-out period of at least one month. According to randomization ,patients will be provided with either Diabeloop system or the usual system.

Patients will be trained for the use of blood glucose meter, of external Insulin Pump and Diabeloop system.

In both treatment periods, the same blood glucose meter will be used throughout the duration of the study.

In two centers (Centre Hospitalier Sud-Francilien and Grenoble), a pre-study will be performed during four weeks to improve the efficacy of Diabeloop system with data collection, to test the manual settings by health care providers and patients and to check the good-working of the follow-up platform.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetic patient for at least two years
* Patient treated by external insulin pump for at least 6 months
* Patient with HbA1c ≤ 10%; dosage of less than 4 months done in analysis laboratory medical or equivalent.
* Patient requiring a daily dose of insulin ≤ 50 units
* Patient domiciled in an area with Global System for Mobile Communication (GSM)
* Not isolated patient, not living alone, or having a person "resource" living nearby and having a phone and the key of its place of residence
* Patient not envisaging a journey outside France during the "closed-loop" period
* Patient aged over 18 years
* Patient affiliated to Social Security
* Patient who agreed to participate in the study and who signed an informed consent

Exclusion Criteria:

* Patient with any serious illness that may impair study participation
* Patient having a treatment known to have a significant interference on the glycemia.
* Patient enjoying a measure of legal protection
* Pregnant woman or likely to be

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2017-03-30 (Actual); Primary Completion 2018-08-28 (Actual); Study Completion 2018-08-28 (Actual)

PRIMARY OUTCOMES:
Percentage of time spent in the tight glycemic control area 70-180 mg/dl continuously measured for 12 weeks | For 12 weeks
  measurement of glucose by CGM

SECONDARY OUTCOMES:
Percentage of time spent in the glycemic range 70-180 mg/dl, 80-140 mg/dl and in blood glucose >180 mg/dL during nights and during 24 hours for 12 weeks | During 24 hours for 12 weeks
  measurement of glucose by CGM
Measurement of HbA1c at the onset and at the end of each period of treatment | During 12 weeks for each period of treatment
  Dosage of HbA1c every 3 months
Average blood glucose levels throughout the full period | During 12 weeks for each period of treatment
  measurement of glucose by CGM
Calculated risks of hypo- and hyperglycemia (LBGI, HBGI) throughout the full period during 12 weeks | Throughout the full period during 12 weeks
  measurement of glucose by CGM
Total supplies of insulin during tests | During 12 weeks for each period
  total basal and bolus by 24h
Number of hyper-glycemic events defined by American Diabetes Association (ADA) : severe hyperglycemia > 360 mg/dl (20 mmol/l) measured by CGM or significant ketose (acetonemia > 3 mmol/l) | During 12 weeks for each period
  measurement of glucose by CGM
Number of hypoglycemic events, defined by any threshold crossing 60 mg/dl ( 3,33 mmol/l); 70 mg/dl (3,9 mmol/l) and < 54 mg/dl (3 mmol/l) measured by the CGM | During 12 weeks for each period
  measurement of glucose by CGM
Measuring the oral carbohydrates intake during the last week of each period of treatment | During 24 hours for one week before the end of each period of treatment
  data collected on a booklet
Number of technical problems causing interruptions of the closed loop | During 12 weeks for the closed loop period
  technical incidents data collected during the study
Percentage of time spent in good-working mode during the closed loop period | During 12 weeks for the closed loop period
  measurement of glucose by CGM
For the use and the acceptance, a satisfaction survey will be done on the daily management of diabetes, the modification of daily life with the system dan the fear of hypoglycemia | During 12 weeks at the end of each period of treatment
  DTSQ satisfaction questionnaire, with scale from 6 to 0 where 0 is the worth and 6 the best outcome.
Percentage of time spent in blood glucose <70 mg/dl continuously measured for 12 weeks | For 12 weeks
  measurement of glucose by CGM

CONTACTS AND LOCATIONS:
Locations (12):
- France (12):
  - Centre Hospitalier Universitaire Jean Minjoz, Besançon
  - Centre Hospitalier Universitaire, Caen
  - Centre Hospitalier Sud-Francilien, Corbeil-Essonnes
  - Centre Hospitalier Universitaire, Grenoble
  - Centre Hospitalier Universitaire, Lyon
  - Centre Hospitalier Universitaire, Marseille
  - Centre Hospitalier Universitaire, Montpellier
  - Centre Hospitalier Universitaire, Nancy
  - Centre Hospitalier Universitaire, Nantes
  - Centre Hospitalier Universitaire, Reims
  - Centre Hospitalier Universitaire, Strasbourg
  - Centre Hospitalier Universitaire, Toulouse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Benhamou PY, Adenis A, Tourki Y, Pou S, Madrolle S, Franc S, Kariyawasam D, Beltrand J, Klonoff DC, Charpentier G. Efficacy of a Hybrid Closed-Loop Solution in Patients With Excessive Time in Hypoglycaemia: A Post Hoc Analysis of Trials With DBLG1 System. J Diabetes Sci Technol. 2024 Mar;18(2):372-379. doi: 10.1177/19322968221128565. Epub 2022 Sep 29. PMID 36172702
- [Derived] Benhamou PY, Franc S, Reznik Y, Thivolet C, Schaepelynck P, Renard E, Guerci B, Chaillous L, Lukas-Croisier C, Jeandidier N, Hanaire H, Borot S, Doron M, Jallon P, Xhaard I, Melki V, Meyer L, Delemer B, Guillouche M, Schoumacker-Ley L, Farret A, Raccah D, Lablanche S, Joubert M, Penfornis A, Charpentier G; DIABELOOP WP7 Trial Investigators. Closed-loop insulin delivery in adults with type 1 diabetes in real-life conditions: a 12-week multicentre, open-label randomised controlled crossover trial. Lancet Digit Health. 2019 May;1(1):e17-e25. doi: 10.1016/S2589-7500(19)30003-2. Epub 2019 May 2. PMID 33323237
- [Derived] Benhamou PY, Madrolle S, Lablanche S, Gallegos A, Tourki Y, Franc S, Doron M, Charpentier G. Comment on Leelarathna et al. Duration of Hybrid Closed-Loop Insulin Therapy to Achieve Representative Glycemic Outcomes in Adults With Type 1 Diabetes. Diabetes Care 2020;43:e38-e39. Diabetes Care. 2020 Oct;43(10):e167. doi: 10.2337/dc20-1291. No abstract available. PMID 32958628
- [Derived] Benhamou PY, Huneker E, Franc S, Doron M, Charpentier G; Diabeloop Consortium. Customization of home closed-loop insulin delivery in adult patients with type 1 diabetes, assisted with structured remote monitoring: the pilot WP7 Diabeloop study. Acta Diabetol. 2018 Jun;55(6):549-556. doi: 10.1007/s00592-018-1123-1. Epub 2018 Mar 9. PMID 29520615